CLINICAL TRIAL: NCT00643708
Title: Transvaginal Ultrasound-Guided Ovarian Interstitial Laser Treatment in Anovulatory Women With Polycystic Ovarian Syndrome: A Randomized Prospective Study on the Effect of Laser Dose Used on the Outcome
Brief Title: Ovarian Laser Treatment in Women With Polycystic Ovarian Syndrome: A Randomized Study on the Laser Dose
Status: Completed | Type: Observational
Sponsor: Shen-Zhen City Maternity and Child Healthcare Hospital (Other)
Responsible Party: Wen-Jie Zhu, Shen-Zhen City Maternity and Child Healthcare Hospital
Other Study IDs: 200602070
Record Dates: First submitted 2008-03-11; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Anovulation; Polycystic Ovary Syndrome; Infertility
Keywords: anovulation; laser; ovarian interstitial; polycystic ovary syndrome; ultrasound-guided
MeSH Terms: conditions — Anovulation; Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- A: 14 cases
  Interventions: Procedure: ovarian interstitial laser treatment
- B: 14 cases
  Interventions: Procedure: ovarian interstitial laser treatment
- C: 14 cases
  Interventions: Procedure: ovarian interstitial laser treatment
- D: 14 Cases
  Interventions: Procedure: ovarian interstitial laser treatment

INTERVENTIONS:
Procedure: ovarian interstitial laser treatment — Different dose of laser: group A, one point per ovary.
  Other Names: Different ovarian laser coagulation points
  Groups: A
Procedure: ovarian interstitial laser treatment — Different dose of laser: group B, two points per ovary.
  Other Names: Different ovarian laser coagulation points
  Groups: B
Procedure: ovarian interstitial laser treatment — Different dose of laser: group c, three points per ovary.
  Other Names: Different ovarian laser coagulation points
  Groups: C
Procedure: ovarian interstitial laser treatment — Different dose of laser: group D, four-five points per ovary.
  Other Names: Different ovarian laser coagulation points
  Groups: D

SUMMARY:
BACKGROUND: A new effective way, transvaginal ultrasound-guided ovarian interstitial laser-coagulation treatment, in management of anovulation in patients with polycystic ovary syndrome (PCOS), has been presented in the data published. But, the optimal number of laser coagulation points in the ovarian interstitial to be applied at the procedure is unclear. This clinic trial aims to explore an optimal laser dose for this new protocol. METHODS: Fifty-six PCOS women with clomifene citrate-resistant underwent ultrasound-guided transvaginal ovarian interstitial YAG-laser treatment. By random list table，all subjects were randomly divided into four groups in terms of the number of laser coagulation points made in their ovaries as follows: group A, one coagulation point per ovary; group B, two points; group C, three points; group D, four to five points. The size of each point was about 10 mm in diameter on the ovarian plane monitored by transvaginal ultrasound. Postoperative ovulation rate, pregnancy rate and some biochemical parameters were compared among four groups.

DETAILED DESCRIPTION:
Materials and methods Subject selection Fifty-six patients with anovulatory infertility due to PCOS were included in the study between January 2005 and December 2007. All women presented with oligo-/amenorrhea and anovulation for at least 2 years and were seeking pregnancy. The mean (± SD) age was 29.1 ± 3.1 years and the mean duration of infertility 3.3 ± 2.0 years. The mean body mass index (BMI) was 22.9 ± 3.5 kg/m2. All subjects had polycystic ovaries on transvaginal ultrasound scan (TVS) (Aloka-1000, UST-985, 5 MHz transvaginal probe, Aloka Co. Ltd, Tokyo, Japan), and the diagnosis of PCOS was made according to criteria of The Rotterdam (The Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group, 2003). Serum concentrations of FSH (5.4±2.3 IU/L), LH (11.8±3.2IU/L) and T (3.79±1.54nmol/L) were assessed at the third day of progesterone-induced bleeding (natural progesterone injection; Guangzhou Minxing pharmaceutical company, Guang-Zhou, China). TVS examination revealed bilateral ovarian enlargement and 10-30 subcapsular follicles of 2-8 mm in diameter in unilateral ovary with a stromal hypertrophy. All cases have received incremental clomifene citrate (CC) doses (50, 100, and 150mg), to which they failed to respond. A normal hysterosalpingography or laparoscopy had to have been recorded in the past three years prior to ovarian interstitial laser treatment. Any contraindications to surgery, previous treatment with LOD and the presence of tubal or male factors for infertility were considered as exclusion criteria. The study was approved by the Ethics Committee of Shen-Zhen Maternity and Child Healthcare Hospital and the Institutional Review Board of Shen-Zhen Bureau of Science and Technology of China. Subjects all signed an informed consent form.

Protocol Study design This was a prospective, randomized study. Fifty-six subjects meeting the enrolled criteria were randomly divided into four groups of A、B、C、D according to a computer-generated random list. Randomization occurred after patients agreed to inclusion in the study (Figure 1). After randomization, women who were allocated in same group were intervened with same laser dosage during ovarian interstitial laser treatment. For each group of A、B、C、D, the number of laser coagulation points made in their ovaries as follows: group A, one coagulation point per ovary; group B, two points; group C, three points; group D, four to five points. To each point, the size of laser coagulation zone was 10 mm in diameter (a light spot of diameter 10 mm on the ovarian plane monitored by transvaginal ultrasound).

Techniques of ovarian interstitial laser treatment The procedure of transvaginal ultrasound-guided ovarian interstitial laser treatment has been detailed in previous data (Zhu et al., 2006). All participants were treated on the third day after progesterone-induced menstruation period. An intramuscular injection of 50-100mg of Pethidine (Pethidine Hydrochloride Injection, Shenyang First Pharmaceutical, NEPG, Shen-Yang, China) was administered to each women about 30 minutes before starting the operation. After emptying their bladder, the women were placed in lithotomy. They were then prepared using an aseptic vulva and vaginal douche. TVS was performed and the widest ovarian plane was found. Usually, one to three intraovarian points can be predetermined in the widest ovarian plane, in other words, one to three laser coagulation points can be accomplished on the widest ovarian plane. If not, the next largest ovarian plane was chosen as the next option until three to five laser coagulation points have be made in unilateral ovary. For each treatment point, a fibre optic cable of 400 um in diameter was sent to intraovarian point by means of a 17-gauge, 35-cm-long needle (K-OPS-1035-Cook IVF; Brisbane, Australia) and the electrical laser (XH-YAG-100 Laser; Wuhan Xinghua Photoelectricity Co. Ltd, Wu-Han, China) was activated persistently for two to five minutes with a power of 3-5 W and current of 8-10 A, until a 10-mm light spot appeared on the ovarian plane. In group A, only one laser treatment point was made per ovary; and group B, two points; group C, three points; group D, four to five points. The women stayed in bed for two to three hours after the surgery, after which they were re-examined with TVS in order to rule out intra-abdominal haemorrhage prior to discharge.

Postoperative Monitoring Serum hormone concentrations At the second, fourth and sixth month after the operation, a blood sample was taken on day three of menstrual cycle for measurement of serum levels of LH, FSH, testosterone, prolactin (PRL), estradiol (E2) and progesterone if the women had a regular ovulation and menstrual cycle. If not, the blood sample was taken on day three of progesterone-induced withdrawal bleeding. Another blood sample was taken on day 21 of the same cycle in order to measure the serum concentration of progesterone when ovulation could not be diagnosed by TVS.

Follicle development and ovulation Follicular growth and ovulation was monitored monthly by TVS at four to five days intervals after the operation. The scanning was repeated after two to three days when the leading follicle reached diameter of 12 mm. When the dominant follicles reached a diameter of 16 mm. LH surge was detected by urinalysis. Combined this result with TVS, ovulation and the timing of sexual intercourse could be confirmed. If the ovulation intervals during the six postoperative months were within a range of 21-35 days, the woman was documented as a responder having regular ovulation. If spontaneous ovulation and menstruation did not occur during six postoperative months, the woman was categorized as a nonresponder. The women whose status was between both would be categorized as having irregular ovulation.

Pregnancy and miscarriage A urine pregnancy test was performed if spontaneous menstruation did not occur during 16-19 days following ovulation. The pregnancy rate was calculated based on the women who conceived. Miscarriage would be considered, if gestational sac without cardiac action or previous cardiac action stopped, although a urine pregnancy test was positive.

Adverse effects Adverse effects, including intra-abdominal haemorrhage, infection, injuries of internal organs and failure of ovarian function, were recorded.

Analysis of the data Women were divided into four groups according to the number of laser coagulation points made in their ovarian interstitial as follows: group A (n=14) treated with one laser coagulation point per ovary, group B (n=14) two points, group C (n=14) three points, group D (n=14) four to five points. The means ± SD of the baseline and postoperative second, fourth and sixth month values among the four groups were calculated for the serum LH, FSH, testosterone, PRL, progesterone, E2 levels. Analysis of variance was used for statistical analysis. The ovulation rate and pregnancy rate were calculated based on the cases of postoperative spontaneous ovulation and pregnancy. Contingency table analysis was used to compare success rates, with P<0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. anovulatory women with clomifene citrate (CC)-resistant polycystic ovary syndrome(PCOS)
2. A normal hysterosalpingography or laparoscopy had to have been recorded
3. infertility

Exclusion Criteria:

1. Any contraindications to surgery
2. previous treatment with LOD
3. presence of tubal or male factors for infertility

Ages: 23 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifty-six patients with anovulatory infertility due to PCOS were included in the study between January 2005 and December 2007. All women presented with oligo-/amenorrhea and anovulation for at least 2 years and were seeking pregnancy. The mean (± SD) age was 29.1 ± 3.1 years and the mean duration of infertility 3.3 ± 2.0 years. The mean body mass index (BMI) was 22.9 ± 3.5 kg/m2. All subjects had polycystic ovaries on transvaginal ultrasound scan (TVS) (Aloka-1000, UST-985, 5 MHz transvaginal probe, Aloka Co. Ltd, Tokyo, Japan), and the diagnosis of PCOS was made according to criteria of The Rotterdam (The Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group, 2003).
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Serum hormone concentrations,Follicle development and ovulation,Pregnancy and miscarriage | 2 months

SECONDARY OUTCOMES:
Serum hormone concentrations,Follicle development and ovulation,Pregnancy and miscarriage,Adverse effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jie Zhu, Master, Study Chair — Shen-Zhen City Maternity and Child Healthcare Hospital

REFERENCES:
- [Derived] Zhu W, Chen M, Fu Z, Li X, Qin C, Tang X, Chen X. Repeat transvaginal ultrasound-guided ovarian interstitial laser treatment improved the anovulatory status in women with polycystic ovarian syndrome. Eur J Obstet Gynecol Reprod Biol. 2012 May;162(1):50-4. doi: 10.1016/j.ejogrb.2012.02.008. Epub 2012 Mar 6. PMID 22397748